CLINICAL TRIAL: NCT05904717
Title: A Phase 2a, Multi Centre, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Effect of 12 Weeks Treatment With Oral PXS-4728A on Microglia Activation, as Measured by Positron Emission Tomography, in Participants With Isolated Rapid Eye Movement Sleep Behavior Disorder
Brief Title: Effect of PXS-4728A on Microglia Activation in Participants With Isolated Rapid Eye Movement Sleep Behaviour Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PXS4728A-IRBD-201
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: REM Sleep Behavior Disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (PXS-4728) (Experimental): IP Name: PXS-4728 Dosage: 15 mg Mode: oral administration (PO)
  Interventions: Drug: PXS-4728 (A)
- B (Matching Placebo) (Placebo Comparator): Matching placebo to PXS-4728
  Interventions: Drug: Matching Placebo (B)

INTERVENTIONS:
Drug: PXS-4728 (A) — Participants will receive once daily (QD) for period of 12 weeks
  Arms: A (PXS-4728)
Drug: Matching Placebo (B) — Participants will receive once daily (QD) for period of 12 weeks
  Arms: B (Matching Placebo)

SUMMARY:
This study is to investigate the safety and efficacy of PXS-4728A as an intervention therapy in participants with iRBD. This study will be conducted in participants aged 50 to 80 years of age and will investigate a single dose level.

DETAILED DESCRIPTION:
Up to 48 participants are planned to be screened and approximately 40 participants are planned to be enrolled in this study. Participants will be randomized to receive either active IP or matching placebo in a ratio of 3:1 (30 active and 10 placebo).

Study participation will consist of a Screening period of up to 2 weeks to confirm participant eligibility. Once confirmed as eligible, participants will be able to enroll in the study and will be required to attend the clinical site on Day 1 for treatment assignment, initial dosing, and Baseline assessments.

Oversight of the study will be provided by a Data Safety Monitoring Committee (DSMC) comprising the Principal Investigator (PI), the local Medical Monitor (MM), and a representative of the Sponsor, at a minimum.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent in accordance with GCP, International Council for Harmonisation (ICH) and local regulations.
2. Male or female aged 50 to 80 (inclusive) as of the date of Baseline visit.
3. Clinical diagnosis of iRBD according to International Classification of Sleep Disorders (ICSD)-3 criteria.
4. Objective evidence of 1 or more features of parkinsonism, impaired olfaction and/or impaired color vision discrimination, which have been associated with an increased risk for transitioning to a synucleinopathy in the opinion of the Investigator.
5. Screening PET scan demonstrates robust PK11195 signal in striato-cortical region of interest in the opinion of the Investigator.
6. Liver Function Tests (LFTs): alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN); total bilirubin ≤ 1.5 × ULN; serum albumin ≥ 2.8 g/dL.
7. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (human chorionic gonadotropin [hCG]) at Screening. WOCBP who engage in heterosexual intercourse and men whose sexual partners are WOCBP must agree to use highly effective, double barrier contraception during the study and for a period of 90 days following final dosing. Double barrier contraception is defined as a condom and 1 other form of the following:

   1. Contraceptive pill
   2. Depot or injectable birth control
   3. Intrauterine Device (IUD)
   4. Contraceptive skin implant, (eg, Implanon NXT®)
   5. Hormonal vaginal ring, (eg, NuvaRing®)
   6. Documented evidence of surgical sterilization at least 6 months prior to the Screening visit, (ie, bilateral tubal ligation, oophorectomy, salpingectomy, or total hysterectomy for women or vasectomy for men).

   Must be willing to remain on their current form of contraception for the duration of the study.

   Note: For participants with same-sex partners or who are otherwise abstinent from heterosexual intercourse, total abstinence (defined as abstinence from penile-vaginal intercourse), when this is the preferred and usual lifestyle of participants, may be considered an acceptable form of contraception.
8. Women not of childbearing potential must be postmenopausal for ≥ 12 months. Postmenopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrheic female participants. Willing and able to have the types of diagnostic procedures required by the protocol, such as neuroimaging, phlebotomy, and other testing.
9. Willing and able to take oral drug therapy according to the study protocol.
10. Willing and able to undertake radiological scans (PET, MRI) and utilize smartphone apps/ devices to complete assessments.

Exclusion Criteria:

1. Meets diagnostic criteria for a degenerative neurologic disorder such as Parkinson's disease, Multiple System Atrophy, Dementia with Lewy Bodies, etc.
2. Screening PET scan does not demonstrate robust PK11195 signal in striato-cortical region of interest in the opinion of the Investigator.
3. RBD associated with narcolepsy.
4. Dementia (Mild Cognitive Impairment permitted).
5. Unstable medications (stable use [minimum 4 weeks] allowed for treatment of affective symptoms [mood disorders] and dream enactment [eg, melatonin, clonazepam, etc]).
6. Untreated or uncontrolled severe obstructive sleep apnea (OSA).
7. Females who are pregnant or breastfeeding.
8. Body mass index (BMI) > 35.0 kg/m2.
9. Any known hypersensitivity to the IP, radioligand or their constituents.
10. Serious neurological disorder, such as uncontrolled epilepsy or stroke.
11. History of psychotic symptoms requiring antipsychotic treatment or exposure to typical or atypical antipsychotics or other dopamine blocking agents within 6 months prior to Screening.
12. History of suicidal attempt/s or ideation/s within the prior 6 months.
13. Gastrointestinal conditions that may affect the absorption of IP (eg, ulcerative colitis, gastric bypass, or active duodenal or gastric ulcers).
14. History of significant medical event/s within 6 months prior to the Screening visit, at the discretion of the PI. This includes, but is not limited to, a cerebrovascular event or a myocardial infarction.
15. Any significant uncontrolled cardiac arrhythmia, including but not limited to second and third degree atrioventricular (AV) block.
16. History of head trauma with loss of consciousness for more than 5 minutes within the past 6 months.
17. Use of drugs historically associated with liver injury, hepatic steatosis, or steatohepatitis in the 4 weeks prior to Screening.
18. History of liver cirrhosis (fibrosis stage 4), or hepatic decompensation (eg, ascites, hepatic encephalopathy, variceal bleeding, etc.) or history of other forms of chronic liver disease (for example Hepatitis B, Hepatitis C, autoimmune liver disease, primary biliary sclerosis, primary sclerosing cholangitis, Wilsons disease, hemochromatosis, A1At deficiency, history of liver transplantation).
19. Active known chronic or relevant acute infections, such as HIV (Human Immunodeficiency Virus), viral hepatitis, or tuberculosis. Participants with a positive test result may participate in the study, at the discretion of the Investigator, if further diagnostic analysis (according to local practice/guidelines) establishes conclusively that the participant has no evidence of active infection.
20. Solid liver lesions other than hemangiomas.
21. Suspicion or diagnosis or history of hepatocellular carcinoma (HCC).
22. Sustained supine hypertension ≥ 180 mmHg systolic or 110 mmHg diastolic, exceeding levels defined by local guidelines ie, ≥ 140/90 mmHg per UK standards. Sustained is defined as the average of 3 observations, each at least 10 minutes apart, with the participant having been supine and at rest for at least 5 minutes prior to each measurement. Uncontrolled cases of elevated BP, based on PI discretion, will be discussed on a case-by-case basis with the Sponsor in consultation with the MM and PI.
23. History of symptomatic orthostatic hypotension (OH) which interferes with the participant's day to day level of functioning. OH is defined as a decrease of ≥ 20 mmHg systolic or ≥ 10 mmHg diastolic when changing from supine to standing position, after having been in supine position for at least 5 minutes.
24. Current unstable angina.
25. Congestive heart failure (New York Heart Association [NYHA] Class 3 or 4).
26. Heart rate ≤ 50 beats per minute (bpm) as tested on 3 occasions, 10 minutes apart.
27. Abnormal 12-lead ECG results, which in the opinion of the Investigator will prevent participation in the study.
28. Uncontrolled diabetes defined as an HbA1c ≥ 9.5% in the 3 months prior to or at Screening.
29. Prior diagnosis of cancer and evidence of continued malignancy within the past 3 years (with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or in situ prostate cancer with normal prostate-specific antigens post resection).
30. Any major surgical procedure within 30 days prior to the Screening visit. Minor surgery is per the discretion of the Investigator.
31. Severely impaired renal function with creatinine clearance < 30 mL/min.
32. Active alcohol or substance use disorder within the past 12 months, at the discretion of the Investigator.
33. Depression of moderate severity or more on the Patient Health Questionnaire (PHQ-9) ≥ 10 at Screening. Note: participants with scores ≥ 10 due to indications in Questions 3 (sleep), 4 (tiredness), and/or 7 (concentration), with no clinical signs of depression, can be included at the discretion of the Investigator following discussion with the Sponsor and MM.
34. Participants with clinically significant abnormalities (as determined by the Investigator) in clinical laboratory tests at Screening, as assessed by the study-specific clinical laboratory. A single repeat test may be conducted if deemed necessary.
35. Participation in any trial of a device (including, but not limited to transcranial magnetic stimulation [TMS], near-infrared [NIR], and red-light therapy [λ = 600-1070 nm]), investigational medicinal product, supplement, surgical treatment, cognitive/behavioral therapy, physiotherapy, or active exercise study within 30 days (or 5 half-lives of an investigational medicinal product, whichever is longer) prior to Screening.
36. Any reason which would impede the ability to safely undertake radiological scans (PET, MRI) such as metal implants, claustrophobia, inability to lie still in the scanner for the scanning period etc.
37. Chronic inflammatory or autoimmune disorder.
38. Receipt of any live vaccine within 4 weeks or any vaccine within 2 weeks prior to Screening.
39. Regular use of anti-inflammatory/immunomodulating medications including prednisolone or other oral steroids (within 3 months of Screening), non-steroidal anti inflammatories including high dose aspirin (> 75 mg), diclofenac, and meloxicam (within 2 weeks of Screening), and immunosuppressant drugs including mycophenolate, methotrexate, rituximab, cyclophosphamide, and alemtuzumab (within 6 months of Screening).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
To assess the reduction of microglial activation across striato-cortical regions | Up to Week 12
  Measured by translocator protein (TSPO) positron emission tomography (PET) imaging.
To assess the safety and tolerability of PXS-4728A as determined by adverse events (AEs) | Up to Week 24
  AEs will be coded using the most recent version of MedDRA®

SECONDARY OUTCOMES:
To assess the reduction of microglial activation across the whole brain and cortical and subcortical regions of interest (ROIs) | Up to Week 12
  Measured by translocator protein (TSPO) positron emission tomography (PET) imaging.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Parkinsons Disease Research Clinic - Macquarie University, Macquarie, New South Wales
  - Cognitive Neuroscience Brain & Mind Centre, Camperdown, Sydney
- Clinical Neuroscience Nuffield Department of Clinical Neurosciences, Oxford, United Kingdom